CLINICAL TRIAL: NCT05334693
Title: Immunotherapy With ex Vivo Expanded Haploidentical Natural Killer Cells as Consolidation Strategy for Children/Young Adults With AML
Brief Title: Expanded Haploidentical Natural Killer Cells as Consolidation Strategy for Children/Young Adults With AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Belarusian Research Center for Pediatric Oncology, Hematology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HaploNK_consolidation_AML
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Natural killer cells; Immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expanded haploidentical NK cell immunotherapy (Experimental): After a lymphodepleting chemotherapy a patient receive two intravenous infusions of expanded haploidentical NK cells.
  Interventions: Biological: Expanded haploidentical NK cells

INTERVENTIONS:
Biological: Expanded haploidentical NK cells — Two doses of expanded haploidentical NK cells (30-100 x 10^6 cells /kg).

SUMMARY:
The purpose of this study is to estimate the efficacy of immunotherapy with ex vivo expanded haploidentical NK cells as consolidation therapy for children/young adults with intermediate risk AML.

DETAILED DESCRIPTION:
Immunotherapy with NK cells may improve the treatment results in AML. For better efficiency high cell doses or several infusions of NK cells are required. For this purpose, donor NK cells are expanded in the presence of feeder K562-mbIL21-41BBL cell line. The cycle of immunotherapy includes chemotherapy (cyclophosphamide, fludarabine) followed by two doses of NK cells infusion.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* primary intermediate risk AML in molecular complete remission;
* primary high risk AML in molecular complete remission awaiting unrelated HSCT;
* Karnofsky or Lansky performance scale greater or equal to 70;
* written informed consent.

Donors:

* haploidentical family donor;
* donor suitable for cell donation and apheresis according to standard criteria;
* written informed consent.

Exclusion Criteria:

Patients:

* uncontrolled infection;
* severe hepatic dysfunction: SGOT or SCPT >=5x upper limit of normal for age;
* positive serology for human immunodeficiency virus (HIV).

Donors:

* pregnancy;
* positive serology for HIV, hepatitis B or C.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | 2 years
  Time from achievement of CR to the time of relapse or death from any cause.
Overall survival (OS) | 2 years
  The proportion of patients with overall survival

SECONDARY OUTCOMES:
Persistence of donor NK cells | 21 days after the first infusion
  Days of persistence of donor NK cells
Number of T, B, NK, activated T and NK cells after immunotherapy | 28 days after the first infusion
  Analysis of T, B, NK, activated T and NK cells numbers (cells/microL) after NK infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Aleinikova, MD, Prof, Principal Investigator — Belarussian Research Center for Pediatric Oncology, Hematology and Immunology
Locations (1):
- Belarussian Research Center for Pediatric Oncology, Hematology and Immunology, Minsk, Minsk Oblast, Belarus